CLINICAL TRIAL: NCT00138177
Title: A Phase I Study of Suberoylanilide Hydroxamic Acid (Vorinostat) in Combination With 5-Fluorouracil, Leucovorin, and Oxaliplatin (mFOLFOX) in Patients With Colorectal Cancer and Other Solid Tumors
Brief Title: Suberoylanilide Hydroxamic Acid, Fluorouracil, Leucovorin, and Oxaliplatin in Treating Patients With Progressive Metastatic or Unresectable Colorectal Cancer or Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00083; NCI-2009-00083 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000439445; I 55305 (Other: Roswell Park Cancer Institute); 6789 (Other: CTEP)
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage III Colon Cancer; Stage III Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Vorinostat; Fluorouracil

ARMS (1):
- Treatment (vorinostat, mFOLFOX) (Experimental): Patients receive oral SAHA once or twice daily on days 1-3. Patients also receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 4 followed by fluorouracil IV over 46 hours on days 4-5. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 10 patients are treated at the MTD.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Drug: vorinostat; Drug: fluorouracil

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU

SUMMARY:
This phase I trial is studying the side effects and best dose of suberoylanilide hydroxamic acid when given together with fluorouracil, leucovorin, and oxaliplatin in treating patients with progressive metastatic or unresectable colorectal cancer or solid tumor. Drugs used in chemotherapy, such as suberoylanilide hydroxamic acid, fluorouracil, leucovorin, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Suberoylanilide hydroxamic acid may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of suberoylanilide hydroxamic acid when administered with fluorouracil, leucovorin calcium, and oxaliplatin in patients with progressive metastatic or unresectable colorectal cancer or other solid tumors.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this regimen in these patients. II. Determine the pharmacokinetics of oxaliplatin, fluorouracil, and suberoylanilide hydroxamic acid in these patients.

OUTLINE: This is a dose-escalation study of suberoylanilide hydroxamic acid (SAHA).

Patients receive oral SAHA once or twice daily on days 1-3. Patients also receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 4 followed by fluorouracil IV over 46 hours on days 4-5. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 10 patients are treated at the MTD.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer
* Metastatic or unresectable disease OR diagnosis of solid tumor
* No known brain metastases
* ECOG 0-1 OR Karnofsky 70-100%
* Life expectancy > 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST and ALT ≤ 3 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No ongoing or active infection
* No neuropathy > grade 1
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to study drugs
* No psychiatric illness or social situation that would preclude study compliance
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* Prior bevacizumab and/or cetuximab allowed
* No concurrent routine or prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* More than 4 weeks since prior radiotherapy
* Recovered from prior therapy
* At least 2 weeks since prior valproic acid
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-07; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of vorinostat | 2 weeks
  Graded according to the NCI CTCAE.
Grade 3, 4, or 5 adverse events graded using the NCI CTCAE version 4.0 | Up to 30 days after completion of study treatment

SECONDARY OUTCOMES:
Response, evaluated using the new international criteria proposed by the RECIST committee | Up to 4 weeks after completion of study treatment
  To be assigned a status of PR or CR, changes in tumor measurements must be confirmed by repeat assessments that should be performed 4 weeks or more after the criteria for response are first met.
Gene expression studies for evidence of up-regulation or down-regulation, obtained from microarray testing and changes in expression patterns of TS | Up to 4 weeks after completion of study treatment
  Carried out with real time quantitative RT-PCR assays.
Pharmacokinetic analysis for vorinostat and 5-FU | Days 1 and 15
DPD activity | Up to 8 days after the first dose of vorinostat (course 1)
  Tabulated by dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States